CLINICAL TRIAL: NCT01408030
Title: North American Study of Epistaxis in HHT (NOSE)
Brief Title: North American Study of Epistaxis in Hereditary Hemorrhagic Telangiectasia (HHT)
Acronym: NOSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James Gossage (Other)
Collaborators: HHT Foundation International (Unknown)
Responsible Party: Sponsor-Investigator, James Gossage, Director of Pulmonary Vascular Diseases and HHT, Augusta University
Organization: Augusta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GHSU 1008041
Record Dates: First submitted 2011-08-01; First posted 2011-08-02 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic; Epistaxis
Keywords: epistaxis; HHT; bevacizumab; tranexamic acid; nosebleed; estrogen
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — Sodium Chloride; Bevacizumab; Vascular Endothelial Growth Factor A; Estriol; Estrogens; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo spray (Placebo Comparator): sterile saline
  Interventions: Drug: Sterile saline
- Bevacizumab spray (Active Comparator): bevacizumab 1%
  Interventions: Drug: Bevacizumab
- Estriol spray (Active Comparator): Estriol 0.1%
  Interventions: Drug: Estriol
- Tranexamic acid spray (Active Comparator): tranexamic acid 10%
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Sterile saline — 0.9%, 0.1 ml spray in each nostril bid
  Other Names: Saline
  Arms: Placebo spray
Drug: Bevacizumab — 1% solution in saline, 0.1 ml spray in each nostril bid
  Other Names: Avastin; Vascular endothelial growth factor (VEGF) inhibitor
  Arms: Bevacizumab spray
Drug: Estriol — 0.1% suspension in methylcellulose, 0.1 ml spray in each nostril bid
  Other Names: Estrogen
  Arms: Estriol spray
Drug: Tranexamic Acid — 10% solution in saline, 0.1 ml spray in each nostril bid
  Other Names: Lysteda
  Arms: Tranexamic acid spray

SUMMARY:
The purpose of the NOSE Study is to carefully examine the efficacy and safety of 3 nasal sprays (bevacizumab, estriol, and tranexamic acid), compared to placebo, for the treatment of HHT related nosebleeds.

DETAILED DESCRIPTION:
140 patients with moderate to severe epistaxis secondary to HHT will be randomized to receive one of four intranasal sprays for a period of 12 weeks and then followed for an additional 12 weeks off therapy. Enrollment will occur over a period of 18-36 months. The primary endpoint will be the frequency of epistaxis. Secondary endpoints will include duration of epistaxis, the Hoag Epistaxis Severity Score (ESS), a quality of life survey, satisfaction with treatment, hemoglobin and ferritin levels, transfusion requirements, and treatment failure. The sprays will be: saline spray (Placebo); estriol 0.1% in methylcellulose suspension (EST); tranexamic acid 10% in saline (TA), and bevacizumab 1% in saline (BEV). All sprays will be applied to the nasal mucosa by an identical spray bottle at a dose of 0.1 ml per nostril twice daily (total dose of 0.4 ml daily). Thus, the delivered doses will be: EST, 0.4 mg/day; TA, 40 mg/day; BEV, 4 mg/day.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of definite or possible HHT by the Curacao criteria (Shovlin 2000) or a positive DNA test for HHT (as characterized by a disease causing mutation in the gene coding for endoglin, activin like kinase 1, or SMAD-4). According to the Curacao criteria, a definite diagnosis of HHT is defined as having at least 3 of the following criteria while a possible diagnosis is defined as 2 criteria:

   1. Spontaneous and recurrent epistaxis.
   2. Multiple telangiectasias at characteristic sites (lips, oral cavity, fingers, nose).
   3. Visceral lesions such as gastrointestinal telangiectasias and arteriovenous malformations (AVM) in lung, brain, spine and liver.
   4. A history of definite HHT in a first degree relative using these same criteria.
2. Epistaxis of at least 1 minute (on average) and which occurs at least once weekly when averaged during the preceding 8 weeks.
3. Epistaxis severity score (ESS) of at least 3.0.
4. Age of at least 18 years.
5. Written and informed consent obtained prior to study entry.
6. Subject is able and willing to return for outpatient visits.
7. The epistaxis is considered to be clinically stable during the past 8 weeks in the clinical judgment of the investigator (i.e. no major changes in frequency or duration of epistaxis or in transfusion requirements).
8. Negative pregnancy test at enrollment.

Exclusion Criteria:

1. Allergy to any of the active treatment agents or their spray additives.
2. Estimated life expectancy less than 1 year.
3. A psychiatric or substance abuse problem that is expected to interfere with study compliance.
4. History of deep venous thrombosis (DVT), pulmonary embolism (PE), acute myocardial infarction (MI), arterial thromboembolism, or ischemic stroke in the past 6 months.6. History of receiving more than 12 units of red blood cells in the past 12 weeks.

7. Presence of an untreated coagulopathy that is felt to be contributing to the 5. History of estrogen receptor positive breast cancer. epistaxis. 8. Presence of active disseminated intravascular coagulation. 9. Uncontrolled hypertension (systolic BP >160 and/or diastolic BP >100). 10. Presence of untreated brain AVM. 11. Presence of active malignancy in the brain, lung, or colon. 12. Presence of symptomatic heart failure. 13. Use of estrogens, epsilon aminocaproic acid, tranexamic acid, or thalidomide by any route for more than 1 week in the past 12 weeks. Any use of a VEGF inhibitor by any route in the past 24 weeks.

14. Baseline use of the following anticoagulants is not allowed: warfarin or other vitamin K antagonists at any dose; unfractionated or low molecular weight heparins at standard doses for treatment of venous thromboembolism (VTE); or aspirin at >325 mg/day. Baseline use of the following anticoagulants is allowed: heparins at standard doses for VTE prophylaxis; clopidogrel; or aspirin at ≤325 mg/day.

15. Addition of new treatments for epistaxis in the past 12 weeks (including laser ablation of nasal telangiectasias and over the counter medications).

16. Presence of another overt cause (e.g. overt gastrointestinal bleeding) that is felt to be significantly contributing to anemia.

17. Lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Gossage, MD, Principal Investigator — Augusta University
Locations (6):
- United States (6):
  - University of California Los Angeles, Los Angeles, California
  - Georgia Regents University, Augusta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Oregon Health Sciences University, Portland, Oregon
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whitehead KJ, Sautter NB, McWilliams JP, Chakinala MM, Merlo CA, Johnson MH, James M, Everett EM, Clancy MS, Faughnan ME, Oh SP, Olitsky SE, Pyeritz RE, Gossage JR. Effect of Topical Intranasal Therapy on Epistaxis Frequency in Patients With Hereditary Hemorrhagic Telangiectasia: A Randomized Clinical Trial. JAMA. 2016 Sep 6;316(9):943-51. doi: 10.1001/jama.2016.11724. PMID 27599329
- See also: HHT Foundation website — http://www.hht.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the HHT clinics at 6 sites if they met all of the following criteria: age >=18; diagnosis of definite or possible HHT; epistaxis lasting at least 1 minute, occurring at least once weekly, and clinically stable during the preceding 8weeks; and had an Epistaxis Severity Score (ESS) of at least 3.0.
Pre-assignment Details: 123 patients provided consent but 1 withdrew consent and 1 was excluded due to brain arteriovenous malformation. Therefore 121 patients were randomized and included in participant flow. 1 patient in the estriol group was subsequently removed after it was discovered that she was taking estrogen outside the protocol (protocol violation).
Period: Treatment Phase (on Drug)
Arm/Group | Bevacizumab Spray | Estriol Spray | Tranexamic Acid Spray | Placebo Spray
Started | 29 | 31 | 33 | 28
Completed | 26 | 24 | 32 | 25
Not Completed | 3 | 7 | 1 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 2 | 6 | 0 | 3
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Period: Observation Phase (Off Drug)
Arm/Group | Bevacizumab Spray | Estriol Spray | Tranexamic Acid Spray | Placebo Spray
Started | 26 | 24 | 32 | 25
Completed | 22 | 18 | 26 | 21
Not Completed | 4 | 6 | 6 | 4
Not completed — Lost to Follow-up | 0 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 1 | 3
Not completed — Physician Decision | 0 | 1 | 2 | 0
Not completed — Other | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab Spray | Estriol Spray | Tranexamic Acid Spray | Placebo Spray | Total
Number analyzed (Participants) | 29 | 30 | 33 | 28 | 120
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 47.8 [42.8 to 52.9] | 56.6 [52 to 61.2] | 53 [48.2 to 57.8] | 53 [48.6 to 57.3] | 52.8 [39.9 to 65.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 14 | 13 | 52
  Male | 16 | 18 | 19 | 15 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 28 | 30 | 33 | 28 | 119
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Definite HHT [Count of Participants; unit: Participants] | 26 | 29 | 32 | 26 | 113
Epistaxis history [Median (Inter-Quartile Range); unit: bleeding episodes per week] | 10.0 [5.0 to 14.0] | 7.0 [7.0 to 14.0] | 7.8 [5.5 to 14.5] | 7.0 [5.0 to 15.0] | 7.0 [3.0 to 14.0]
Epistaxis severity score [Mean (Full Range); unit: units on a scale] | 5.16 [4.75 to 5.57] | 5.19 [4.71 to 5.68] | 5.43 [4.94 to 5.91] | 5.71 [5.04 to 6.38] | 5.37 [4.71 to 6.38]

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Epistaxis
Description: Bleeding episodes per week
Time Frame: Weeks 5-12 of active treatment phase
Population: Participants were included in this analysis (106) if they had at least 3 weeks of data during weeks 5-12; therefore the number of participants analyzed do not equal the number who finished the active treatment phase (120). 2 patients were lost to follow up, 5 dropped out before week 5, 6 filled out diaries incorrectly, and 1 had no diary.
Measure: Median (Inter-Quartile Range); unit: Bleeding episodes per week
Arm/Group | Bevacizumab Spray | Estriol Spray | Tranexamic Acid Spray | Placebo Spray
Number analyzed (Participants) | 24 | 25 | 30 | 27
Bleeding episodes per week | 7.0 [4.5 to 10.5] | 8.0 [4.0 to 12.0] | 7.5 [3.0 to 11.0] | 8.0 [3.0 to 14.0]
Statistical Analysis 1: Comparison: Bevacizumab Spray vs Estriol Spray vs Tranexamic Acid Spray vs Placebo Spray; Test type: Other — Two sided testing was performed with a significance level of 0.05; p = 0.97, ANOVA

2. Secondary Outcome: Duration of Epistaxis
Description: Total minutes of bleeding per week
Time Frame: 5-12 weeks of active treatment
Population: Participants were included in this analysis (112) if they had at least 3 weeks of data during weeks 5-12; therefore the number of participants analyzed do not equal the number who finished the active treatment phase (120). 2 patients were lost to follow up, 5 dropped out before week 5, and 1 had no epistaxis diary.
Measure: Median (Inter-Quartile Range); unit: Total minutes of bleeding per week
Arm/Group | Bevacizumab Spray | Estriol Spray | Tranexamic Acid Spray | Placebo Spray
Number analyzed (Participants) | 26 | 26 | 32 | 28
Total minutes of bleeding per week | 23.5 [13 to 40] | 36.5 [7 to 70] | 44.5 [13.5 to 87.5] | 46 [10 to 84]
Statistical Analysis 1: Comparison: Bevacizumab Spray vs Estriol Spray vs Tranexamic Acid Spray vs Placebo Spray; Test type: Other — Two sided testing was performed with a significance level of 0.05; p = .47, ANOVA

3. Secondary Outcome: Hoag Epistaxis Severity Score
Description: Hoag Epistaxis Severity Score (ESS) is based on 6 nosebleed variables such as frequency and duration which are entered by patients. The ESS has a minimum value of 0 and maximum value of 10, with 10 representing more severe epistaxis.
Time Frame: 12 weeks
Population: Participants were included in this analysis if they completed week 12 (phase 1) and filled out an ESS score. 1 participant each from the bevacizumab and placebo group did not fill out an ESS score at week 12.
Measure: Median (95% Confidence Interval); unit: units on a scale (0-10)
Arm/Group | Bevacizumab Spray | Estriol Spray | Tranexamic Acid Spray | Placebo Spray
Number analyzed (Participants) | 25 | 24 | 32 | 24
units on a scale (0-10) | 3.54 [3 to 4.08] | 3.56 [2.81 to 4.3] | 4.06 [3.5 to 4.61] | 3.74 [3.17 to 4.31]
Statistical Analysis 1: Comparison: Bevacizumab Spray vs Estriol Spray vs Tranexamic Acid Spray vs Placebo Spray; Test type: Other — Two sided testing was performed with a significance level of 0.05; p < 0.001, Mixed Models Analysis — A mixed-model repeated-measures ANOVA was used to analyze ESS for drug and time (baseline, week 12) effects. Listed P value is for time effect; Clinical site and patient were included in the model as random effects

4. Secondary Outcome: Hemoglobin Level
Description: grams/100 ml, assessed at week 12
Time Frame: 12 weeks
Population: 8 participants who finished the active treatment phase did not have a hemoglobin level measured, and thus only 99 were analyzed.
Measure: Median (Inter-Quartile Range); unit: gram/100 ml
Arm/Group | Bevacizumab Spray | Estriol Spray | Tranexamic Acid Spray | Placebo Spray
Number analyzed (Participants) | 23 | 22 | 31 | 23
gram/100 ml | 12.8 [11.7 to 14.1] | 13.1 [12.3 to 14.9] | 11.4 [10 to 13.6] | 13.8 [12.6 to 14.9]
Statistical Analysis 1: Comparison: Bevacizumab Spray vs Estriol Spray vs Tranexamic Acid Spray vs Placebo Spray; Test type: Other — Two sided testing was performed with a significance level of 0.05; p = 0.43, ANCOVA; Adjusted for baseline values and random effect of clinic site

5. Secondary Outcome: Number of Participants Requiring Red Blood Cell (RBC) Transfusion
Description: Number of participants requiring RBC transfusion during weeks 1-12
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Spray | Estriol Spray | Tranexamic Acid Spray | Placebo Spray
Number analyzed (Participants) | 29 | 30 | 33 | 28
Participants | 1 | 2 | 5 | 3
Statistical Analysis 1: Comparison: Bevacizumab Spray vs Estriol Spray vs Tranexamic Acid Spray; Test type: Other — Two sided testing was performed with a significance level of 0.05; p = 0.42, Fisher Exact

6. Secondary Outcome: Number of Participants With Treatment Failure
Description: Treatment failure is defined as the occurrence of one or more of the following during the study: need for nasal surgery or chemical cautery or other new treatment modality to control epistaxis; transfusion of more than 12 units of RBC; severe complications such as acute myocardial infarction, venous thromboembolism, brain hemorrhage; or death
Time Frame: Baseline through 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Spray | Estriol Spray | Tranexamic Acid Spray | Placebo Spray
Number analyzed (Participants) | 29 | 30 | 33 | 28
Participants | 2 | 5 | 0 | 3
Statistical Analysis 1: Comparison: Bevacizumab Spray vs Estriol Spray vs Tranexamic Acid Spray vs Placebo Spray; Test type: Other — Two sided testing was performed with a significance level of 0.05; p = 0.08, Fisher Exact

ADVERSE EVENTS:
Time Frame: Weeks 1-24
Description: Patients were queried at various time points about a specific list of key adverse events and asked for any additional side effects that they may have experienced. Nasal symptoms included rhinorrhea, congestion and sneezing but were not monitored in such a way to allow distinction. Nausea and vomiting were not monitored in such a way to allow distinction and are reported collectively as nausea/vomiting.
Arm/Group | Bevacizumab Spray | Estriol Spray | Tranexamic Acid Spray | Placebo Spray
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30 | 0/33 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/33 | 0/28
Other Adverse Events (participants affected / at risk) | 24/29 | 25/30 | 26/33 | 23/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Spray (N=29) | Estriol Spray (N=30) | Tranexamic Acid Spray (N=33) | Placebo Spray (N=28)
Nasal symptoms (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 12 (12) | 10 (10) | 10 (10) — New symptoms such as congestion and rhinorrhea; excludes nosebleeds
Headache (Nervous system disorders) | 10 (10) | 12 (12) | 10 (10) | 6 (6)
Nausea/vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 10 (10) | 8 (8)
Abdomial pain (Gastrointestinal disorders) | 5 (5) | 2 (2) | 10 (10) | 1 (1)
Vision problem (Eye disorders) | 2 (2) | 2 (2) | 5 (5) | 1 (1)

LIMITATIONS AND CAVEATS:
1. One key limitation is the lack of a baseline epistaxis diary. 2. Drug absorption may have been hampered because of local scab and crust formation causing a barrier to drug penetration. 3. Saline may not be a true placebo due to hydration effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No